CLINICAL TRIAL: NCT04610866
Title: Evaluation of the Safety,Tolerability, Pharmacokinetics, and Pharmacodynamics of Long-term Mitapivat Dosing in Subjects With Stable Sickle Cell Disease: An Extension of a Phase I Pilot Study of Mitapivat
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Long-term Mitapivat Dosing in Subjects With Stable Sickle Cell Disease: An Extension of a Phase I Pilot Study of Mitapivat
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10000049; 000049-H
Record Dates: First submitted 2020-10-30; First posted 2020-11-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-16

CONDITIONS: Sickle Cell Disease; Hemolytic Anemia
Keywords: HbS polymerization; pyruvate kinase; 2,3- diphosphoglycerate; ATP in red blood cells; Hemolytic Anemia
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia, Hemolytic | interventions — mitapivat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Subjects will be treated with a maintenance dose of mitapivat previously assessed for safety and tolerability in the Phase I study for an initial 48 weeks and undergo safety monitoring, evaluation of pharmacokinetics and pharmacodynamics, and assessment of secondary laboratory and clinical endpoints at pre-specified intervals during the study period.
  Interventions: Drug: Mitapivat

INTERVENTIONS:
Drug: Mitapivat — Investigational drug mitapivat (also known as AG-348, AGI-1480 and AGX-0841) is an orally bioavailable, broad-spectrum allosteric activator of alleles of the RBC-specific form of pyruvate kinase (PKR), as well as liver-type pyruvate kinase (PKL) and muscle pyruvate kinase (PKM1 and PKM2).

SUMMARY:
Background:

Sickle cell disease (SCD) is a disorder that causes episodes of acute pain and progressive organ damage. Ways to manage SCD have evolved slowly. Treatments do not always work. Researchers want to see if a drug called mitapivat can help people with SCD.

Objective:

To test the long-term tolerability and safety of mitapivat (or AG-348) in people with SCD.

Eligibility:

Adults age 18-70 with SCD who took part in and benefited from NIH study #19H0097.

Design:

Participants will be screened with a medical history and physical exam. They will give a blood sample. They will have an electrocardiogram to test heart function.

Participants will repeat some of the screening tests during the study.

Participants will complete 6-minute walk tests to measure mobility and function. They will have transthoracic echocardiograms to measure heart and lung function. They will have dual-energy X-ray absorptiometry scans to measure bone health. They will complete online questionnaires that measure their overall health and well-being.

Participants will take the study drug in the form of a tablet twice a day.

Participants will keep a study diary. They will record any symptoms they may have.

Participation will last for about 54 weeks. After 48 weeks, participants can either keep taking the study drug for 48 more weeks or be tapered off of the study drug to complete the study. Those who are on the study for 1 year will have 10 study visits. Those who are on the study for 2 years will have 14 study visits.

DETAILED DESCRIPTION:
Study Description:

The objective of this extension study is to evaluate the safety and tolerability of mitapivat (AG-348) as long-term maintenance therapy for subjects with sickle cell disease (SCD) who have completed the Phase I dose escalation study of mitapivat (NCT04000165, protocol 19H0097). Subjects will be treated with a maintenance dose of mitapivat previously assessed for safety and tolerability in the Phase I study for an initial 48 weeks and undergo safety monitoring, evaluation of pharmacokinetics and pharmacodynamics, and assessment of secondary clinical endpoints at regular intervals over the study period. Exploratory endpoints will allow for investigation of the mechanisms by which mitapivat may modulate red cell metabolism and survival and lead to clinical benefits in SCD. Subjects benefiting from the study drug will have the option to continue therapy for an additional years.

Objectives:

Primary Objective:

- To assess the long-term safety and tolerability of mitapivat in subjects with stable sickle cell disease.

Secondary Objectives:

* To evaluate the pharmacokinetic/pharmacodynamic profile of long-term dosing of mitapivat, as well as its mechanisms of action on the glycolytic pathway in SCD subjects.
* To evaluate hemoglobin (Hb) response, changes in hemolytic markers, functional status, cardiopulmonary function, and health-related quality of life in SCD subjects maintained on mitapivat long-term.
* To monitor SCD-related safety endpoints in SCD subjects maintained on mitapivat long-term.

Tertiary/Exploratory Objectives:

- To assess the feasibility and usability of digital health technology in a drug trial for patients with SCD.

Endpoints:

Primary Endpoints:

- Frequency and severity of AEs and changes in clinical and laboratory parameters over 8 years of therapy with mitapivat.

Secondary Endpoints:

* Change from baseline in pharmacokinetic and pharmacodynamic measures over time.
* Hemoglobin (Hb) response and changes in hemolytic markers at 24 and 48 weeks on mitapivat.
* Sustained Hb response from weeks 12-48.
* Change from baseline in functional and cardiopulmonary status at 24 and 48 weeks on mitapivat.
* Change from baseline in quality of life at 24 and 48 weeks on mitapivat.
* Frequency of acute vaso-occlusive clinical events at 24 and 48 weeks on mitapivat.

Tertiary/Exploratory Endpoints:

- Usability of SCD Warrior digital Microhealth application (app) by providers and participants through simple feedback tools at each protocol visit reviewing ease of use and patient satisfaction.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects completing Study 19H0097 will first be screened for eligibility. Eligibility criteria are identical with the exception of criteria 5.1.4, 5.2.2, and 5.2.3.p. If any of the 15 subjects completing the 19H0097 study are unable to participate in or complete the current extension study (defined as completing 24 weeks of treatment with study drug to allow for assessment of the primary endpoint), then additional new subjects naive to mitapivat treatment may be enrolled to replace them.

Subjects will enroll onto the study and undergo screening. Subjects who do not meet any of the following criteria during screening will not receive the study intervention but will be counted toward study accrual. Screen failures may be rescreened at a later time.

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1.1 Have provided signed written informed consent prior to performing any study procedure, including screening procedures.

1.2 Age between 18-70 years

1.3 Unequivocal diagnosis of HbSS confirmed by hemoglobin electrophoresis performed on patients at least 90 days after a blood transfusion if previously transfused, or DNA genotyping

1.4 No transfusion in the 12 weeks prior to signing consent, or absence of Hb A on hemoglobin analysis (by high-performance liquid chromatography; HPLC)

1.5 Have adequate organ function, as defined by:

1. Serum aspartate aminotransferase (AST) <=2.5 x Upper Limit of Normal (ULN) (unless the increased AST is assessed by the Investigator as due to hemolysis) and alanine aminotransferase (ALT) <=2.5 x ULN.
2. Serum creatinine <=1.25 x ULN. If serum creatinine is >1.25 x ULN, then glomerular filtration rate (based on creatinine) must be >=60 mL/min.
3. Absolute neutrophil count >=1.0 x 10^9/L.
4. Hemoglobin >= 7 g/dL
5. Platelet count >=100 x 10^9/L.
6. Activated partial thromboplastin time and international normalized ratio <=1.5 x ULN, unless the subject is receiving therapeutic anticoagulants.

1.6 For women of reproductive potential, have a negative serum pregnancy test during the screening period. Women of reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy, or tubal occlusion; or who have not been naturally postmenopausal (i.e., who have not menstruated at all for at least the preceding 1 year prior to signing informed consent unrelated to hormonal contraception).

1.7 For women of reproductive potential be abstinent as part of their usual lifestyle, or agree to use one highly effective form of contraception from the time of giving informed consent, during the study, and for 28 days following the last dose of study treatment. Furthermore, due to the potential for mitapivat to reduce the effectiveness of hormonal contraceptives, women using hormonal contraception as a highly effective method of contraception must also utilize an acceptable barrier method while enrolled in the study and for at least 28 days after their last dose of mitapivat. Women using nonhormonal methods of contraception as a highly effective method do not need to use an additional barrier method.

1.8 Be willing to comply with all study procedures for the duration of the study.

EXCLUSION CRITERIA:

2.1 Documented pyruvate kinase deficiency

2.2 Screening hemoglobin level of >= 11 g/dL

2.3 Have a significant medical condition that confers an unacceptable risk to participating in the study, and/or that could confound the interpretation of the study data. Such significant medical conditions include, but are not limited to the following:

1. Poorly controlled hypertension (defined as systolic blood pressure [BP] >150 mmHg or diastolic BP >90 mmHg) refractory to medical management.
2. History of recent (within 24 weeks prior to signing consent) decompensated congestive heart failure; myocardial infarction or unstable angina pectoris; hemorrhagic, embolic, or thrombotic stroke; deep venous thrombosis; or pulmonary or arterial embolism.
3. Cardiac dysrhythmias judged as clinically significant by the Investigator.
4. Heart-rate corrected QT interval-Fredericia's method (QTcF) >480 msec with the exception of subjects with right or left bundle branch block.
5. Clinically symptomatic cholelithiasis or cholecystitis. Prior cholecystectomy is not exclusionary. Subjects with symptomatic cholelithiasis or cholecystitis may be rescreened once the disorder has been treated and clinical symptoms have resolved.
6. History of drug-induced cholestatic hepatitis.
7. Iron overload sufficiently severe to result in a clinical diagnosis by the Investigator of cardiac (e.g., clinically significant impaired left ventricular ejection fraction), hepatic (e.g., fibrosis, cirrhosis), or pancreatic (e.g., diabetes) dysfunction.
8. Have a diagnosis of any other congenital or acquired blood disorder, or any other hemolytic process as defined by a positive direct antiglobulin test (DAT), except mild allo-immunization as a consequence of transfusion therapy.
9. Positive test for hepatitis B surface antigen or hepatitis C virus (HCV) antibody (Ab) with signs of active hepatitis B or C virus infection. If the subject is positive for HCVAb, a reverse transcriptase-polymerase chain reaction test will be conducted. Subjects with hepatitis C may be rescreened after receiving appropriate hepatitis C treatment.
10. Positive test for human immunodeficiency virus 1 or 2 Ab.
11. Active infection requiring any use of systemic antimicrobial agents (parenteral or oral) or Grade >=3 in severity (per National Cancer Institute Common Terminology Criteria for Adverse Events) within 8 weeks prior to signing consent.
12. Diabetes mellitus judged to be under poor control by the Investigator or requiring >3 antidiabetic agents, including insulin (all insulins are considered 1 agent); use of insulin per se is not exclusionary.
13. History of any primary malignancy, with the exception of: curatively treated nonmelanomatous skin cancer; curatively treated cervical or breast carcinoma in situ; or other primary tumor treated with curative intent, no known active disease present, and no treatment administered during the last 3 years.
14. Current or recent history of psychiatric disorder that, in the opinion of the Investigator or Medical Monitor, could compromise the ability of the subject to cooperate with study visits and procedures.
15. Are currently enrolled in another therapeutic clinical trial involving ongoing therapy with any investigational or marketed product or placebo. SCD subjects on hydroxyurea or L-glutamine will also be considered, provided that they have been on an unchanged dose of hydroxyurea or LGlutamine for 12 weeks prior to signing consent. Use of the newer SCD therapies voxelotor or crizanlizumab will not be permitted on this study, and subjects who have received voxelotor or crizanlizumab in the 12 weeks prior to signing consent will be excluded.
16. Have exposure to any investigational drug (other than the current drug, mitapivat), device, or invasive procedure within 12 weeks prior to signing consent. All non-investigational invasive procedures within 12 weeks of signing consent may be considered as a potential exclusion criteria per the PI s discretion.
17. Have had a prior bone marrow or stem cell transplant.
18. Are currently pregnant or breastfeeding.
19. Are currently receiving products that are strong inhibitors of CYP3A4/5 that have not been stopped for (Bullet)5 days or a time frame equivalent to 5 half-lives (whichever is longer), or strong inducers of CYP3A4 that have not been stopped for (Bullet)28 days or a time frame equivalent to 5 half-lives (whichever is longer), prior to signing consent.
20. Are currently receiving hematopoietic stimulating agents (e.g., erythropoietins, granulocyte colony stimulating factors, thrombopoietins) that have not been stopped for a duration of at least 90 days prior to signing consent.
21. Have a history of allergy to sulfonamides if characterized by acute hemolytic anemia, drug-induced liver injury, anaphylaxis, rash of erythema multiforme type or Stevens-Johnson syndrome, cholestatic hepatitis, or other serious clinical manifestations.
22. Have a history of allergy to mitapivat or its excipients (microcrystalline cellulose, croscarmellose sodium, sodium stearyl fumarate, and mannitol).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure: Long-term safety and tolerability of mitapivat in subjects with stable sickle cell disease | 48 weeks
  Frequency and severity of AEs and changes in clinical and laboratory parameters over 48 weeks of maintenance therapy with mitapivat.

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic | 24 and 48 weeks
  Change from baseline in pharmacokinetic and pharmacodynamic measures over time.
To evaluate hemoglobin (Hb) response, changes in hemolytic markers, functional status, cardiopulmonary function, and health-related quality of life in SCD subjects maintained on mitapivat long-term. | 24 and 48 weeks
  - Hemoglobin (Hb) response and changes in hemolytic markers at 24 and 48 weeks on mitapivat. Sustained Hb response from weeks 12-48. - Change from baseline in functional and cardiopulmonary status at 24 and 48 weeks on mitapivat. - Change from baseline in quality of life at 24 and 48 weeks on mitapivat
To monitor SCD-related safety endpoints in SCD subjects maintained on mitapivat long-term. | 24 and 48 weeks
  - Frequency of acute vaso- occlusive events (acute vaso-occlusive pain crisis, acute chest syndrome, hepatic sequestration, splenic sequestration, and priapism) at 24 and 48 weeks on mitapivat.

CONTACTS AND LOCATIONS:
Overall Officials: Swee Lay Thein, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The team is deciding on the matter.

REFERENCES:
- [Derived] D'Alessandro A, Le K, Lundt M, Li Q, Dunkelberger EB, Cellmer T, Worth AJ, Patil S, Huston C, Grier A, Dzieciatkowska M, Stephenson D, Eaton WA, Thein SL. Functional and multi-omics signatures of mitapivat efficacy upon activation of pyruvate kinase in red blood cells from patients with sickle cell disease. Haematologica. 2024 Aug 1;109(8):2639-2652. doi: 10.3324/haematol.2023.284831. PMID 38450513
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000049-H.html